CLINICAL TRIAL: NCT00096213
Title: A Phase II Surgical Trial Of Intralesional Resection Of Low-Grade Intracompartmental Chondrosarcoma Of Bone
Brief Title: S0344 Intralesional Resection in Treating Patients With Chondrosarcoma of the Bone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); American College of Surgeons (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000390349; U10CA032102 (NIH); S0344 (Other: SWOG); ACOSOG-S0344 (Other: ACOSOG)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Sarcoma
Keywords: chondrosarcoma
MeSH Terms: conditions — Sarcoma; Chondrosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgery (Other): intralesional resection
  Interventions: Procedure: conventional surgery

INTERVENTIONS:
Procedure: conventional surgery — surgery

SUMMARY:
RATIONALE: Intralesional resection is a less invasive type of surgery for chondrosarcoma of the bone and may have fewer side effects and improve recovery.

PURPOSE: This phase II trial is studying how well intralesional resection works in treating patients with low-grade chondrosarcoma of the bone.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the probability of local complications (e.g., fracture, nerve palsy, deep venous thrombosis, unexpected rehospitalization, unanticipated reoperation, or death within 2 years) in patients with suspected low-grade intracompartmental chondrosarcoma of the bone undergoing intralesional resection.
* Determine the 5-year probability of local recurrence and development of metastatic disease in patients undergoing this procedure.
* Determine the impact of musculoskeletal tumor reconstruction on the functional status of patients undergoing this procedure.

OUTLINE: This is a multicenter study.

Patients undergo intralesional resection (curettage with high-speed burr). Patients then receive local adjuvant treatment comprising liquid nitrogen, phenol, alcohol, or argon beam to the excision site. The bone cavity is then filled with either polymethyacrylate cement or a bone graft (allograft or homograft). Patients may also have a metal plate installed at the wound site.

Patients are followed every 3 months for 1 year and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 30-60 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Suspected low-grade intracompartmental chondrosarcoma, as defined by the following criteria:

  * Resorption of prior calcifications (indicated by a change in radiographic appearance over time) AND/OR meets at least 2, but no more than 4, of the following criteria:

    * Permeative appearance of medullary bone, defined as presence of tumor around 3 sides of a trabecula of normal bone
    * Endosteal scalloping, defined as > 50% of adjacent cortical thickness
    * Cortical thickening beyond the thickness of adjacent normal bone
    * Bone expansion, defined as a circumferential increase in diameter of the bone beyond the adjacent normal bone
    * Positive (i.e., increased uptake or "hot") bone scan
* No cortical disruption and/or soft tissue mass by radiography and CT scan (3 mm cuts are optimal) or MRI
* No presumptive axial (spinal) involvement
* No multifocal disease by bone scan

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for this tumor

Chemotherapy

* No prior chemotherapy for this tumor

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for this tumor

Surgery

* No prior surgery for this tumor except biopsy*
* No concurrent intramedullary fixation NOTE: *Biopsy is not required

Other

* No prior investigational anticancer agents for this tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-12; Primary Completion 2006-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Probability of local complications | two years

SECONDARY OUTCOMES:
Probability of local recurrence and development of metastatic disease | 5 years
Impact of musculoskeletal tumor reconstruction on functional status | two years

CONTACTS AND LOCATIONS:
Overall Officials: R. Lor Randall, MD, FACS, Study Chair — University of Utah; Janet S. Biermann, MD, Study Chair — University of Michigan Rogel Cancer Center; Edward Cheng, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (23):
- United States (23):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Akron City Hospital, Akron, Ohio
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington